CLINICAL TRIAL: NCT03576183
Title: Randomized Double-Blinded Pilot Study Confirming A Human Challenge Model Using LSN03-016011/A Expressing LT And CS17 And Investigating The Safety Of VLA1701 (An Investigational Oral Cholera And ETEC (Enterotoxigenic E Coli) (Vaccine)
Brief Title: Study Confirming A Human Challenge Model and Investigating The Safety Of VLA1701
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: Johns Hopkins University (Other); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA1701-201
Record Dates: First submitted 2018-05-15; First posted 2018-07-03 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Enterotoxigenic Escherichia Coli Infection; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLA1701 (Active Comparator): VLA1701 is an investigational oral vaccine against LT-ETEC (Labile Toxin-Enterotoxigenic E coli)
  The vaccine is administered orally in 2 doses about 1 week apart.
  Interventions: Biological: VLA1701; Other: Challenge Strain
- Placebo (Placebo Comparator): The buffer component of VLA1701 will be used as Placebo.
  The vaccine is administered orally in 2 doses about 1 week apart.
  Interventions: Biological: Placebo; Other: Challenge Strain

INTERVENTIONS:
Biological: VLA1701 — VLA1701 is an investigational oral vaccine against LT-ETEC (Labile Toxin-Enterotoxigenic E coli)
  Arms: VLA1701
Biological: Placebo — buffer component of VLA1701
  Arms: Placebo
Other: Challenge Strain — LSN03-016011/A

SUMMARY:
This is a single-center, double-blind, placebo-controlled, Phase II vaccination and challenge study designed to confirm a human challenge model with E. coli strain LSN03-016011/A.

DETAILED DESCRIPTION:
This is a single-center, double-blind, placebo-controlled, Phase II vaccination and challenge study designed to confirm a human challenge model with E. coli strain LSN03-016011/A (LT+ (Labile toxin), ST- (Stable toxin), CS17), as well as collect expanded safety and immunogenicity data.

The study will be carried out in two phases:

Vaccination phase: up to 34 subjects will be randomized 1:1 to receive 2 doses of either VLA1701 or placebo orally. The doses will be given 7 days apart and subjects will be followed as an outpatient for safety.

Challenge Phase: 30 Subjects, out of the 34 subjects, will be challenged.

After challenge, subjects will be monitored for diarrhea and other signs/symptoms of enteric illness by daily medical checks, vital sign determinations, grading and weighing of all stools.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant female subjects aged 18 to <50 years;
2. BMI of 19.0 to 35.0 kg/m2
3. Willingness to participate after informed consent has been obtained from the subject prior to any study related procedures.
4. Completion of a training session and demonstration of comprehension of the protocol procedures and knowledge of ETEC-associated illness by passing a written examination.
5. If subject is of childbearing potential:

   1. Negative pregnancy test at screening with understanding to not become pregnant within 28 days after challenge;
   2. Subject has practiced an effective method of contraception during the 30 days before screening (Visit 0);
   3. Subject agrees to employ adequate birth control measures for the duration of the study.

Exclusion Criteria

1. Participated in research involving investigational product within 30 days before planned date of first vaccination or planned use through Day 44;
2. Any prior exposure to ETEC (including LSN03-016011/A) or cholera occupationally or received LT (Or any mutant forms of LT (e.g., LTR192G, LTR192GL211A), ETEC, or cholera vaccine);
3. Subjects with known abnormal stooling patterns (fewer than 3 per week or more than 3 per day);
4. Known allergies to any component of the vaccine;
5. Subjects with known allergies to more than 1 planned antibiotics:
6. History of diarrhea while traveling in a developing country within the last 3 years;
7. Subjects whose occupation involves handling of ETEC or cholera bacteria;
8. Women who are pregnant or breastfeeding;
9. Significant medical conditions including chronic, immunosuppressive, malignant, or gastrointestinal diseases (e.g. History of Irritable Bowel Syndrome (as defined by the Rome III criteria or medical diagnosis) or gastric ulcer disease) or enteric, pulmonary, cardiac, liver or renal disease. Some medical conditions which are adequately treated and stable may be acceptable in the study (e.g. hypertension);
10. Significant abnormalities in screening lab hematology or serum chemistries;
11. Use of any medication known to effect the immune system (e.g. systemic corticosteroids) within 30 days of vaccination or planned use during active study period (excluding inhaled steroids);
12. Evidence of confirmed infection with HIV, Hepatitis B or Hepatitis C;
13. Subjects with IgA (Immunoglobulin A) deficiency (serum IgA < 7 mg/dl or limit of detection of assay);
14. Regular use of antacids, antidiarrheal, loperamide, bismuth subsalicylate, diphenoxylate or similar medication less than 2 weeks prior to enrolling in the study and through the inpatient portion of the study;
15. Known or suspected alcohol abuse or illicit drug use within the last year, positive urine toxicology for drugs of abuse;
16. Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
17. Persons who are in a dependent relationship with the sponsor, an investigator or other study team members, or the study center.
18. Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Taucher, PhD, Study Director — Valneva Austria GmbH
Locations (1):
- Department of International Health Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talaat KR, Porter CK, Chakraborty S, Feijoo BL, Brubaker J, Adjoodani BM, DeNearing B, Prouty MG, Poole ST, Bourgeois AL, Billingsley M, Sack DA, Eder-Lingelbach S, Taucher C. Validation of a Human Challenge Model Using an LT-Expressing Enterotoxigenic E. coli Strain (LSN03-016011) and Characterization of Potential Amelioration of Disease by an Investigational Oral Vaccine Candidate (VLA1701). Microorganisms. 2024 Apr 3;12(4):727. doi: 10.3390/microorganisms12040727. PMID 38674674

RESULTS

PARTICIPANT FLOW:
Groups:
- VLA1701: VLA1701 is an investigational oral vaccine against LT-ETEC (Labile Toxin-Enterotoxigenic E coli)
  The vaccine is administered orally in 2 doses about 1 week apart.
  VLA1701: VLA1701 is an investigational oral vaccine against LT-ETEC (Labile Toxin-Enterotoxigenic E coli)
  Challenge Strain: LSN03-016011/A
- Placebo: The buffer component of VLA1701 will be used as Placebo.
  The vaccine is administered orally in 2 doses about 1 week apart.
  Placebo: buffer component of VLA1701
  Challenge Strain: LSN03-016011/A
Period: Overall Study
Arm/Group | VLA1701 | Placebo
Started | 17 | 17
Completed | 15 | 16
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Challenge Population = all subjects who received two doses of the vaccine and the challenge dose
Groups:
- Total: Total of all reporting groups
Arm/Group | VLA1701 | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (7.89) | 35.1 (9.09) | 35.1 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 12 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 14 | 11 | 25
  White | 0 | 2 | 2
  American Indian or Alaskan Native | 1 | 0 | 1
  Other: Multi-racial | 0 | 1 | 1
  Other: Latino / Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Moderate to Severe Diarrhea
Description: within 120 hours of challenge with ETEC strain LSN03-016011/A.
Time Frame: 5 days after challenge
Population: Challenge Population = all subjects who received two doses of the vaccine and the challenge dose
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 7 | 11

2. Secondary Outcome: Disease Severity Score After Challenge With ETEC Strain LSN03-016011/ A
Description: ETEC diarrhea disease severity score with a score ranging from 0 (no disease) to 8 (most severe disease) utilizing objective signs, subjective Symptoms and stool output.
Time Frame: 7 days after challenge
Population: Challenge Population = all subjects who received two doses of the vaccine and the challenge dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 2.3 (1.7) | 3.7 (1.9)

3. Secondary Outcome: Percentage of Subjects With Solicited Adverse Events
Description: adverse events covered by the subjects memory card
Time Frame: 7days after each vaccination
Population: Safety Population = all subjects who entered into the study and received at least one vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants
  Diarrhea | 17.6 [6.2 to 41.0] | 11.8 [3.3 to 34.3]
  Fever | 0 [0 to 18.4] | 0 [0 to 18.4]
  Nausea | 5.9 [1.0 to 27.0] | 0 [0 to 18.4]
  Bloating | 5.9 [1.0 to 27.0] | 11.8 [3.3 to 34.3]
  Vomiting | 0 [0 to 18.4] | 0 [0 to 18.4]
  Generalized Myalgia | 0 [0 to 18.4] | 0 [0 to 18.4]
  Arthralgia | 0 [0 to 18.4] | 0 [0 to 18.4]
  Abdominal Pain | 5.9 [1.0 to 27.0] | 5.9 [1.0 to 27.0]
  Abdominal Cramping | 0 [0 to 18.4] | 5.9 [1.0 to 27.0]
  Malaise | 0 [0 to 18.4] | 0 [0 to 18.4]
  Headache | 17.6 [6.2 to 41.0] | 11.8 [3.3 to 34.3]
  Loss of appetite | 5.9 [1.0 to 27.0] | 0 [0 to 18.4]
  Dizziness | 0 [0 to 18.4] | 0 [0 to 18.4]
  Fatique | 0 [0 to 18.4] | 5.9 [1.0 to 27.0]
  Urticaria | 0 [0 to 18.4] | 0 [0 to 18.4]
  Chills | 0 [0 to 18.4] | 11.8 [3.3 to 34.3]
  Rash | 0 [0 to 18.4] | 5.9 [1.0 to 27.0]

4. Secondary Outcome: Percentage of Subjects With Any Adverse Events (AE)
Time Frame: until Month 6
Population: Safety Population = all subjects who entered into the study and received at least one vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants
  any unsolicited AE - prior Challenge | 17.6 [6.2 to 41.0] | 23.5 [9.6 to 47.3]
  any unsolicited AE related - prior Challenge | 11.8 [3.3 to 34.3] | 5.9 [1.0 to 27.0]
  any severe unsolicited AE - prior Challenge | 0 [0 to 18.4] | 0 [0 to 18.4]
  any unsolicited AE lead vacc. withdrawn - prior | 0 [0 to 18.4] | 0 [0 to 18.4]
  any unsolicite AE leading discontinuation - prior | 0 [0 to 18.4] | 0 [0 to 18.4]
  any unsolicited AE - entiry study period | 58.8 [36.0 to 78.4] | 76.5 [52.7 to 90.4]
  any unsolicited AE related - entire study period | 11.8 [3.3 to 34.3] | 5.9 [1.0 to 27.0]
  any severe unsolicited AE - entire study period | 5.9 [1.0 to 27.0] | 23.5 [9.6 to 47.3]
  any unsolicited AE leading discontinuation - study | 0 [0 to 18.4] | 0 [0 to 18.4]

5. Secondary Outcome: Number of Subjects With Serious Adverse Events
Time Frame: until Month 6
Population: Safety Population = all subjects who entered into the study and received at least one vaccination
Measure: Number; unit: participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 17 | 17
participants
  prior Challenge | 0 | 0
  entire study period | 0 | 0

6. Secondary Outcome: Percentage of Subjects With Any IMP (Investigational Medicinal Product) Related Adverse Events
Description: unsolicited events
Time Frame: up to Visit 4 (day of challenge, 23 days post first vaccination)
Population: Safety Population = all subjects who entered into the study and received at least one vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants | 11.8 [3.3 to 34.3] | 5.9 [1.0 to 27.0]

7. Secondary Outcome: Percentage of Subjects With IMP-related Serious Adverse Events
Time Frame: up to Visit 4 (day of challenge, 23 days post first vaccination)
Population: Safety Population = all subjects who entered into the study and received at least one vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA1701 | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants | 0 [0 to 18.4] | 0 [0 to 18.4]

ADVERSE EVENTS:
Time Frame: until Month 6
Description: solicited and unsolicited AEs
Arm/Group | VLA1701 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 10/17 | 13/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA1701 (N=17) | Placebo (N=17)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 5 (6) | 8 (8)
Abdominal Tenderness (Gastrointestinal disorders) | 3 (3) | 6 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Culture stool positive (Investigations) | 3 (3) | 2 (2)
Blood Creatinine increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03576183/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03576183/SAP_003.pdf